CLINICAL TRIAL: NCT06408974
Title: A Comparison Of Intrathecal Ketamine Versus Intravenous Dexamethasone For Postoperative Analgesia In Parturients Undergoing Spinal Anaesthesia For Cesarean Section: A Randomised Trial
Brief Title: Comparison Between Ketamine Intrathecal and iv Dexamethasone for Post Cesarean Analgesia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rokaya Mahmoud Khalifa, resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: comparison
Record Dates: First submitted 2023-11-27; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Post Cesarean Analgesia
MeSH Terms: interventions — Ketamine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): will include 30 patients, will receive intrathecal bupivacaine 10mg , ,2mg morphine.
- Ketamine group (Active Comparator): will include 30 patients, will receive intrathecal bupivacaine 10 mg , ,2 mg morphine, ,1 mg/kg ketamine .
  Interventions: Drug: Ketamine
- Dexamethasone group (Active Comparator): will include 30 patients , will receive intrathecal bupivacaine 10 mg , ,2 mg morphine , intravenous dexamethasone 8mg .
  Interventions: Drug: dexamethasone

INTERVENTIONS:
Drug: Ketamine — . Standard monitoring procedures will include pulse oximetry, electrocardiography, and noninvasive arterial pressure prior to anesthetic induction. All patients will be premedicate antibiotic prophylaxis, according to the hospital's protocol. Anesthesia will be induced with intrathecal bupivacaine 10mg and ,1 mg/kg ketamine added in group A under sterile condition
  Arms: Ketamine group
Drug: dexamethasone — . Standard monitoring procedures will include pulse oximetry, electrocardiography, and noninvasive arterial pressure prior to anesthetic induction. All patients will be premedicate antibiotic prophylaxis, according to the hospital's protocol. Anesthesia will be induced with intrathecal bupivacaine 10mg and iv dexamethasone will be added
  Arms: Dexamethasone group

SUMMARY:
The aim of our study is to compare the postoperative analgesic efficacy of intrathecal ketamine added to bupivacaine to that of intravenous dexamethasone in patients undergoing cesarean section under bupivacaine spinal anesthesia.

DETAILED DESCRIPTION:
Caesarean delivery is associated with postoperative pain that may influence recovery, psychological maternal well-being, and breastfeeding Multimodal analgesic regimen including an intrathecal long-acting opioid, non-steroidal anti-inflammatory drugs, and acetaminophen has been suggested to effectively control postoperative pain after caesarean delivery Intravenous dexamethasone is recommended in elective caesarean delivery to decrease postoperative pain. Several systematic reviews and meta-analyses have examined the efficacy of dexamethasone after caesarean delivery and reported decreased postoperative pain and prolonged time to first analgesia In the same context, a meta-analysis of randomized controlled trials in humans suggests that there may be a benefit to using intrathecal ketamine as an adjunct to bupivacaine to improve postoperative pain after cesarean section . The mechanisms of action of intrathecal ketamine are incompletely understood. One study reports that ketamine's high lipophilicity allows for rapid diffusion into the venous system, namely through the azygos vein.

The following parameters will be monitored intraoperatively every 5 min:

* HR, SBP, DBP, and MAP and SpO2 and documented every 15 min. till the end of surgery.
* Any hemodynamic response to skin incision and to subsequent surgical steps will be documented.
* For maintaining HR or systolic in range of more or less than 20% of baseline intraoperatively, ephedrine and intravenous fluids will be used . No other analgesic will be given intraoperatively.
* primperan 0.1 mg/kg will be given at the end of the procedure to all patients.
* All patients will receive 20 iu of oxytocin more till 40 iu or any ueterotonic drugs ( papal,methylergometrine) if needed .
* Postoperative pain will be assessed using an 11-point (0=no pain and 10=worst pain) numeric rating scale (NRS). NRS for pain at rest and when coughing will be assessed serially at 1, 2, 4, 8, 16 and 24 h after surgery. The assessor and the patients will be unaware of the type of intervention received.
* Time for first analgesic request and NRS at first analgesic request will be recorded. The duration of analgesia will be evaluated as the time from block administration to the time at which patient complained of pain or NRS ≥4 on assessment at serial intervals and nalurphine will be used as rescue analgesia . Total doses of analgesics required in the first 24 h will be recorded.
* The presence of postoperative nausea and vomiting during the first 24 h will be recorded. Postoperative nausea or vomiting will be treated with 0.1 mg/kg of ondansetron. If the patient did not respond to ondansetron, then metoclopramide 10 mg will be given IV. Occurrence of any complications such as sedation ,nystagmus ,dizziness will be assessed

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years
* Body mass index (BMI) of 18-35 kg/m2
* Patients with the American Society of Anesthesiologists (ASA) physical status I/II,
* Patients scheduled for elective cesarean section .
* females. .

Exclusion Criteria:

* Patient refusal
* Allergy to local anaesthetics
* Infection at the site of injection
* Coagulopathy,
* Chronic pain syndromes
* Prolonged opioid medication
* Patients who received any analgesic 24 h before surgery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
first call for analgesia | 24 hours
  The first call for analgesia (the elapsed time from the time of spinal anaesthesia until the first postoperative analgesic use after the end of the surgery, which will be administrated based on patient request).

SECONDARY OUTCOMES:
nausea & vomiting | 24 hours
  Incidence of Postoperative nausea & vomiting (PONV) 24 hours postoperatively.
analgesic requirement | 24 hours
  The total analgesic requirement in 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: nagwa mo ibraheem, prof, Principal Investigator — assuit study

REFERENCES:
- [Result] Gamez BH, Habib AS. Predicting Severity of Acute Pain After Cesarean Delivery: A Narrative Review. Anesth Analg. 2018 May;126(5):1606-1614. doi: 10.1213/ANE.0000000000002658. PMID 29210789
- [Result] Bornstein E, Husk G, Lenchner E, Grunebaum A, Gadomski T, Zottola C, Werner S, Hirsch JS, Chervenak FA. Implementation of a Standardized Post-Cesarean Delivery Order Set with Multimodal Combination Analgesia Reduces Inpatient Opioid Usage. J Clin Med. 2020 Dec 22;10(1):7. doi: 10.3390/jcm10010007. PMID 33375192
- [Result] Heesen M, Rijs K, Hilber N, Eid K, Al-Oweidi A, Rossaint R, Klimek M. Effect of intravenous dexamethasone on postoperative pain after spinal anaesthesia - a systematic review with meta-analysis and trial sequential analysis. Anaesthesia. 2019 Aug;74(8):1047-1056. doi: 10.1111/anae.14666. Epub 2019 May 6. PMID 31058317
- [Result] Sohnen S, Dowling O, Shore-Lesserson L. Single dose perioperative intrathecal ketamine as an adjuvant to intrathecal bupivacaine: A systematic review and meta-analysis of adult human randomized controlled trials. J Clin Anesth. 2021 Oct;73:110331. doi: 10.1016/j.jclinane.2021.110331. Epub 2021 May 5. PMID 33962333
- [Result] Bion JF. Intrathecal ketamine for war surgery. A preliminary study under field conditions. Anaesthesia. 1984 Oct;39(10):1023-8. doi: 10.1111/j.1365-2044.1984.tb08895.x. PMID 6496899
- [Result] Ituk U, Thenuwara K. The effect of a single intraoperative dose of intravenous dexamethasone 8 mg on post-cesarean delivery analgesia: a randomized controlled trial. Int J Obstet Anesth. 2018 Aug;35:57-63. doi: 10.1016/j.ijoa.2018.03.008. Epub 2018 Mar 26. PMID 29773484